CLINICAL TRIAL: NCT02870946
Title: The Effect of Simultaneous Renal Replacement Therapy on Extracorporeal Membrane Oxygenation Support for Cardiogenic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Director of Center for Cardiac Intensive Care, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z161100000516017
Record Dates: First submitted 2016-08-08; First posted 2016-08-17 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Cardiogenic Shock
Keywords: Extracorporeal Membrane Oxygenation; Cardiogenic Shock; Renal Replacement Therapy
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simultaneous RRT (Experimental): The patients in the simultaneous RRT arm will receive RRT when ECMO is commenced.
  Interventions: Procedure: Simultaneous RRT
- Standard care (Experimental): The patients in the standard care arm will not receive RRT when ECMO is commenced. Only when a patient demonstrates AKI and fulfills any one of the criteria of the conventional RRT indication, RRT would be delivered.
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Simultaneous RRT — The patients in the simultaneous RRT arm will receive RRT when ECMO is commenced. (see Study Description)
  Arms: Simultaneous RRT
Procedure: Standard care — The patients in the standard care arm will not receive RRT when ECMO is commenced. Only when a patient demonstrates AKI and fulfills any one of the criteria of the conventional RRT indication, RRT would be delivered.
  Arms: Standard care

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a temporary mechanical circulatory support device for cardiogenic shock (CS) patients. During ECMO support, renal replacement therapy (RRT) facilitate more rapid metabolic or uremic control and more effective prevention and management of fluid overload which happened in critical state. CS patients who are likely to receive ECMO support will be enrolled and randomized with a 1:1 allocation to a simultaneous RRT arm vs. standard care arm.

1. The patients in the simultaneous RRT arm will receive RRT when ECMO is commenced.
2. The patients in the standard care arm will not receive RRT when ECMO is commenced. Only when a patient demonstrates AKI and fulfills any one of the criteria of the conventional RRT indication during ECMO support or after ECMO weaning, conventional-indication RRT would be delivered.

The primary outcome is all-cause 30-day mortality after ECMO is commenced

DETAILED DESCRIPTION:
Background:

Extracorporeal membrane oxygenation (ECMO) is a temporary mechanical circulatory support device for cardiogenic shock (CS) patients. Patients with fluid overload (FO) and sever metabolic disorder in the early phase of ECMO support exhibit higher hospital mortality. Simultaneous renal replacement therapy (RRT) is routinely used to facilitate more rapid metabolic or uremic control and more effective prevention and management of fluid overload when ECMO is commenced in some ECMO centers registered in the Extracorporeal Life Support Organization (ELSO). However, high-quality evidence to support the strategy of simultaneous RRT during ECMO support is currently lacking. The investigators aim to perform a single center, randomized, controlled trial to evaluate the impact of simultaneous RRT on outcomes during ECMO support for CS patients.

Hypotheses:

The investigators hypothesize that simultaneous RRT with ECMO will improve survival, reduce morbidity, and shorten duration on ECMO support, duration on invasive ventilation, total days of ICU stay and hospitalization, and time to recovery from electrolyte disturbance.

Design:

Prospective, single-center, randomized, open-label trial comparing simultaneous RRT and standard care strategies in terms of overall survival.

CS patients who are likely to receive ECMO support will be enrolled and randomized with a 1:1 allocation to a simultaneous RRT arm vs. standard care arm.

1. Simultaneous RRT arm: The continuous renal replacement therapy (CRRT) machine is primed and connected to the patient by a "machine in-line" CRRT access after randomization. The drainage tube of the CRRT machine is connected to the ECMO circuit where is after the membrane lung, and the return tube before the membrane lung. The simultaneous RRT begins after ECMO is commenced and finishes when a patient has been weaned from ECMO. If a patient has AKI (The definition is described in outcomes.) after ECMO weaning and fulfills any of the criteria of the following conventional indications, conventional-indication RRT should be delivered with independent CRRT access with a central venous catheter: (1) Serum potassium≥6.0 mmol/L, (2) Serum bicarbonate≤10 mmol/L, or (3) urine output < 0.5 ml/kg/h for 24 hours after ECMO weaning.
2. Standard care arm: Only when a patient demonstrates AKI and fulfills any one of the criteria of the conventional indication mentioned above during ECMO support or after ECMO weaning, conventional-indication RRT should be delivered. The "machine in-line" CRRT access or independent CRRT access is separately used when RRT is delivered during ECMO support or after ECMO weaning.

Primary outcome:

All-cause 30-day mortality after ECMO is commenced.

Secondary outcomes:

Morbidity (acute kidney injury, infection), duration on ECMO support, duration on invasive ventilation, total days of ICU stay and hospitalization, and time to recovery from electrolyte disturbance.

Number of subjects required:

The baseline hospital mortality (66%) of CS patients with ECMO support was obtained from the investigators' previous study. Based on their literature research, early initiation of RRT could reduce the mortality by 18%. Assuming all-cause 30-day mortalities in the control and intervention groups of 66% and 48%, respectively, with a two-sided significance of 0.05 and a power of 0.8, a total of 262 patients (131 for each arm) will be required, including an estimated dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 70 years.
2. Admission to ICU.
3. Criteria for the diagnosis of CS as follows: (1) systolic blood pressure less than 90 mmHg for 30 min, a mean arterial pressure less than 65 mmHg for 30 min, or vasopressors required to achieve a blood pressure ≥ 90 mmHg; (2) pulmonary congestion or elevated left-ventricular filling pressures; and (3) signs of impaired organ perfusion with at least one of the following criteria: (a) altered mental status; (b) cold, clammy skin; (c) oliguria; and (d) increased serum lactate.
4. ECMO will supply cardiopulmonary support to the patient.

Exclusion Criteria:

1. Refusal of consent.
2. Received or decided to receive RRT before ECMO was commenced.
3. Fulfilled the criteria for Chronic Kidney Disease (either of the following present for >3 months): (1) Albuminuria (albumin excretion rate > 30 mg/24 hours; albumin-to-creatinine ratio > 30 mg/g); (2) urine sediment abnormalities; (3) electrolyte and other abnormalities due to tubular disorders; (4) abnormalities detected by histology; (5) structural abnormalities detected by imaging; and (6) history of kidney transplantation.
4. Received ECMO bridging to a long-term ventricle assist device or heart transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days

SECONDARY OUTCOMES:
Rate of acute kidney injury | 30 days
  AKI is defined as any of the following: (1) increase in serum creatinine (SCr) by ≥ 26.5lmol/l in 48 hours; (2) increase in SCr to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or (3) urine output < 0.5 ml/kg/h for 6 hours (urine output is only assessed when the CRRT machine is absent or with a fluid removal rate of 0 ml/h).
Rate of infection | 30 days
  Any kinds of infection
Duration on ECMO support | 60 days
Rate of successful weaning from ECMO | 30 days
Duration on invasive ventilation | 60 days
ICU length of stay | 60 days
Hospital length of stay | 60 days
Time to recovery from electrolyte and metabolic disturbance | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No